CLINICAL TRIAL: NCT05246514
Title: An Open-label, Single-arm, Phase 2 Study to Evaluate the Efficacy and Safety of Trastuzumab Deruxtecan (T-DXd) for Patients With HER2-mutant Metastatic NSCLC Who Have Disease Progression on or After at Least One-line of Treatment (DESTINY-Lung05)
Brief Title: A Single Arm Phase 2 Study to Evaluate Efficacy and Safety of Trastuzumab Deruxtecan for Patients With HER2 Mutant NSCLC
Acronym: DL-05
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7811C00001
Record Dates: First submitted 2022-02-11; First posted 2022-02-18 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: HER2-mutant Non-Small Cell Lung Cancer
Keywords: DL05; T-DXd; HER2-mutant Non-Small Cell Lung Cancer; NSCLC; Trastuzumab deruxtecan; ERBB2
MeSH Terms: interventions — trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- T-DXd arm (Experimental): Participants will receive T-DXd as an IV infusion Q3W, on Day 1 of each 3-week cycle.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — administered as an IV infusion
  Other Names: T-DXd, DS-8201a

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of T-DXd in participants with HER2 mutant metastatic non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented metastatic non-squamous NSCLC.
* Has relapsed from or is refractory to at least one-line of anticancer treatment.
* Documented HER2 exon 19 or 20 mutation from central FFPE tumour tissue testing.
* WHO or ECOG performance status of 0 or 1.
* Presence of at least one measurable lesion assessed by the investigator based on RECIST 1.1.
* LVEF ≥ 50% within 28 days before enrolment.

Exclusion Criteria:

* Mixed small cell lung cancer, squamous histology NSCLC, and sarcomatoid histology variant NSCLC.
* Corrected QT interval (QTcF) prolongation to > 470 ms (females) or > 450 ms (males), based on average of the screening triplicate 12-lead ECG.
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Has unresolved toxicities from previous anticancer therapy, defined as toxicities (excluding alopecia) not yet resolved to Grade ≤1 or baseline. Participants with clinically stable chronic Grade 2 toxicity not reasonably expected to be exacerbated by study intervention may be included only after consultation with the AstraZeneca study physician or designee.
* Has been previously treated with HER2-targeted therapies, except for pan-HER class TKIs or has received prior treatment with an ADC which consists of an exatecan derivative that is a topoisomerase I inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-09-23 (Actual); Study Completion 2026-03-16 (Estimated)

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Research Site, Baoding
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Linyi
  - Research Site, Nanjing
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yangzhou
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7811C00001&attachmentIdentifier=4aca569e-8f50-4761-90f5-52f8b9212e55&fileName=d7811c00001-csp-v2_sign-off_version_Redacted_PDFA.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7811C00001&attachmentIdentifier=68e28558-1517-42b2-8680-e6d7c9bbccec&fileName=d7811c00001-sap-ed-2_8Aug2024_Redacted_PDFA.pdf&versionIdentifier=
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7811C00001&attachmentIdentifier=71ebc875-bf50-46e2-8717-039305429672&fileName=D7811C00001_-___Primary_Clinical_Study_Report_Synopsis_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | T-DXd Arm
Started | 72
Completed | 0
Not Completed | 72
Not completed — Ongoing in the study at data cut-off date | 58
Not completed — Withdrawal by Subject | 1
Not completed — Death | 13

BASELINE CHARACTERISTICS:
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: Years] | 57.0 [34 to 76]
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 72
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 72
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: ICR-assessed ORR (Objective Response Rate)
Description: Confirmed ORR, defined as the percentage of participants with confirmed complete response or partial response, as assessed by independent central review(ICR) based on RECIST 1.1.
Time Frame: At an average of approximately 14 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Percentage of participants | 58.3 [46.1 to 69.8]

2. Secondary Outcome: Investigator-assessed ORR (Objective Response Rate)
Description: Confirmed ORR is defined as the percentage of participants who have a confirmed CR or confirmed PR, as determined by the investigator at local site per RECIST 1.1
Time Frame: An average of approximately 14 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Percentage of participants | 58.3 [46.1 to 69.8]

3. Secondary Outcome: ICR-assessed and Investigator-assessed DoR (Duration of Response)
Description: DoR is time from the initial confirmed response (CR or PR) until documented tumour progression or death from any cause.
Time Frame: At an average of approximately 14 months
Population: Full analysis set (patients with confirmed objective response included in the analysis)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Months
  ICR-assessed | NA [6.1 to NA] — NA - Not calculated, estimate cannot be calculated as the median time frame was not reached. Insufficient number of participants with events for median and upper limit of 95% confidence interval.
  Investigator-assessed | 9.0 [7.2 to NA] — NA - Not calculated, estimate cannot be calculated. Insufficient number of participants with events for upper limit of 95% confidence interval.

4. Secondary Outcome: ICR-assessed and Investigator-assessed DCR (Disease Control Rate)
Description: DCR is the percentage of participants who achieved confirmed CR, PR, or SD during study intervention.
Time Frame: Approximately 6 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Percentage of participants
  ICR-assessed | 91.7 [82.7 to 96.9]
  Investigator-assessed | 93.1 [84.5 to 97.7]

5. Secondary Outcome: ICR-assessed and Investigator-assessed PFS (Progression-free Survival)
Description: PFS is the time from date of enrolment until first objective radiographic tumour progression or death from any cause.
Time Frame: An average of approximately 14 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Months
  ICR-assessed | NA [7.2 to NA] — NA - Not calculated, estimate cannot be calculated as the median PFS time was not reached. Insufficient number of participants with events for median and upper limit of 95% confidence interval.
  Investigator-assessed | 10.8 [7.2 to NA] — NA - Not calculated, estimate cannot be calculated. Insufficient number of participants with events for upper limit of 95% confidence interval.

6. Secondary Outcome: OS (Overall Survival)
Description: OS is the time from date of enrolment until death from any cause.
Time Frame: An average of approximately 22 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Months | NA [NA to NA] — NA - Not calculated, estimate cannot be calculated as the median OS was not reached. Insufficient number of participants with events for median and lower and upper limits of 95% confidence interval.

7. Secondary Outcome: ICR-assessed CNS-PFS (Central Nervous System Progression-free Survival)
Description: CNS-PFS is the time from date of enrolment until CNS tumour progression per RECIST 1.1 as assessed by ICR due to any cause in the absence of CNS progression.
Time Frame: An average of approximately 14 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
Months | NA [7.8 to NA] — NA - Not calculated, estimate cannot be calculated as the median CNS-PFS was not reached. Insufficient number of participants with events for median and upper limit of 95% confidence interval.

8. Secondary Outcome: Serum Concentrations of T-DXd
Description: Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for T-DXd.
Time Frame: An average of approximately 14 months
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
μg/mL
  Cycle 1 Pre-dose: number analyzed (Participants) | 71
  Cycle 1 Pre-dose | NA (NA) — NA - Not calculated, estimate cannot be calculated as too many values were below the lower limit of quantification.
  Cycle 1 End of infusion: number analyzed (Participants) | 71
  Cycle 1 End of infusion | 120.5 (18.33)
  Cycle 1 5 hour post-dose: number analyzed (Participants) | 71
  Cycle 1 5 hour post-dose | 106.1 (77.96)
  Cycle 2 Pre-dose: number analyzed (Participants) | 69
  Cycle 2 Pre-dose | 3.072 (121.6)
  Cycle 2 End of infusion: number analyzed (Participants) | 70
  Cycle 2 End of infusion | 117.4 (18.79)
  Cycle 3 Pre-dose: number analyzed (Participants) | 64
  Cycle 3 Pre-dose | 5.262 (111.2)
  Cycle 3 End of infusion: number analyzed (Participants) | 64
  Cycle 3 End of infusion | 120.9 (17.04)
  Cycle 4 Pre-dose: number analyzed (Participants) | 61
  Cycle 4 Pre-dose | 8.014 (60.69)
  Cycle 4 End of infusion: number analyzed (Participants) | 61
  Cycle 4 End of infusion | 118.4 (18.44)
  Cycle 6 Pre-dose: number analyzed (Participants) | 55
  Cycle 6 Pre-dose | 9.046 (67.91)
  Cycle 8 Pre-dose: number analyzed (Participants) | 44
  Cycle 8 Pre-dose | 10.05 (68.29)

9. Secondary Outcome: Serum Concentrations of Total Anti-HER2 Antibody
Description: Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for total anti-HER2 antibody.
Time Frame: An average of approximately 14 months
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
ug/mL
  Cycle 1 Pre-dose: number analyzed (Participants) | 71
  Cycle 1 Pre-dose | NA (NA) — NA - Not calculated, estimate cannot be calculated as too many values were below the lower limit of quantification.
  Cycle 1 End of infusion: number analyzed (Participants) | 71
  Cycle 1 End of infusion | 127.5 (21.93)
  Cycle 1 5 hour post-dose: number analyzed (Participants) | 71
  Cycle 1 5 hour post-dose | 118.0 (18.85)
  Cycle 2 Pre-dose: number analyzed (Participants) | 69
  Cycle 2 Pre-dose | 2.866 (148.7)
  Cycle 2 End of infusion: number analyzed (Participants) | 70
  Cycle 2 End of infusion | 120.1 (39.66)
  Cycle 3 Pre-dose: number analyzed (Participants) | 64
  Cycle 3 Pre-dose | 4.582 (126.4)
  Cycle 3 End of infusion: number analyzed (Participants) | 64
  Cycle 3 End of infusion | 125.9 (16.87)
  Cycle 4 Pre-dose: number analyzed (Participants) | 61
  Cycle 4 Pre-dose | 6.974 (84.38)
  Cycle 4 End of infusion: number analyzed (Participants) | 61
  Cycle 4 End of infusion | 121.3 (16.80)
  Cycle 6 Pre-dose: number analyzed (Participants) | 55
  Cycle 6 Pre-dose | 8.083 (95.47)
  Cycle 8 Pre-dose: number analyzed (Participants) | 44
  Cycle 8 Pre-dose | 9.193 (87.45)

10. Secondary Outcome: Serum Concentrations of DXd
Description: Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for DXd.
Time Frame: An average of approximately 14 months
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | T-DXd Arm
Number analyzed (Participants) | 72
ng/mL
  Cycle 1 Pre-dose: number analyzed (Participants) | 71
  Cycle 1 Pre-dose | NA (NA) — NA - Not calculated, estimate cannot be calculated as too many values were below the lower limit of quantification.
  Cycle 1 End of infusion: number analyzed (Participants) | 71
  Cycle 1 End of infusion | 5.384 (47.55)
  Cycle 1 5 hour post-dose: number analyzed (Participants) | 71
  Cycle 1 5 hour post-dose | 12.90 (69.38)
  Cycle 2 Pre-dose: number analyzed (Participants) | 69
  Cycle 2 Pre-dose | 0.1751 (119.4)
  Cycle 2 End of infusion: number analyzed (Participants) | 70
  Cycle 2 End of infusion | 2.657 (70.96)
  Cycle 3 Pre-dose: number analyzed (Participants) | 64
  Cycle 3 Pre-dose | 0.2423 (110.6)
  Cycle 3 End of infusion: number analyzed (Participants) | 64
  Cycle 3 End of infusion | 2.310 (50.12)
  Cycle 4 Pre-dose: number analyzed (Participants) | 61
  Cycle 4 Pre-dose | 0.3226 (53.71)
  Cycle 4 End of infusion: number analyzed (Participants) | 61
  Cycle 4 End of infusion | 2.139 (51.35)
  Cycle 6 Pre-dose: number analyzed (Participants) | 55
  Cycle 6 Pre-dose | 0.3295 (58.92)
  Cycle 8 Pre-dose: number analyzed (Participants) | 44
  Cycle 8 Pre-dose | 0.3714 (57.45)

ADVERSE EVENTS:
Time Frame: An average of approximately 16 months
Arm/Group | T-DXd Arm
All-Cause Mortality (participants affected / at risk) | 13/72
Serious Adverse Events (participants affected / at risk) | 33/72
Other Adverse Events (participants affected / at risk) | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd Arm (N=72)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Death (General disorders) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Covid-19 (Infections and infestations) | 5 (5)
Covid-19 pneumonia (Infections and infestations) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 6 (7)
Ascites (Gastrointestinal disorders) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-DXd Arm (N=72)
Vomiting (Gastrointestinal disorders) | 23 (49)
Asthenia (General disorders) | 11 (28)
Fatigue (General disorders) | 8 (12)
Influenza like illness (General disorders) | 5 (5)
Malaise (General disorders) | 6 (9)
Pyrexia (General disorders) | 4 (4)
Covid-19 (Infections and infestations) | 26 (29)
Covid-19 pneumonia (Infections and infestations) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 41 (77)
Pneumonia (Infections and infestations) | 10 (10)
Alanine aminotransferase increased (Investigations) | 29 (48)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 5 (9)
Aspartate aminotransferase increased (Investigations) | 41 (77)
Bile acids increased (Investigations) | 5 (10)
Abdominal distension (Gastrointestinal disorders) | 9 (18)
Bilirubin conjugated increased (Investigations) | 5 (6)
Blood alkaline phosphatase increased (Investigations) | 12 (17)
Blood bilirubin increased (Investigations) | 8 (10)
Blood creatinine increased (Investigations) | 5 (6)
Blood lactate dehydrogenase increased (Investigations) | 8 (10)
Gamma-glutamyltransferase increased (Investigations) | 18 (24)
Lymphocyte count decreased (Investigations) | 16 (36)
Neutrophil count decreased (Investigations) | 46 (163)
Platelet count decreased (Investigations) | 39 (81)
Weight decreased (Investigations) | 11 (14)
Abdominal pain upper (Gastrointestinal disorders) | 6 (12)
Weight increased (Investigations) | 5 (6)
White blood cell count decreased (Investigations) | 47 (191)
Decreased appetite (Metabolism and nutrition disorders) | 30 (50)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (10)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 (14)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (18)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 (37)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (27)
Hypochloraemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 16 (26)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (19)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (5)
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 (9)
Insomnia (Psychiatric disorders) | 8 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 16 (26)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Hypertension (Vascular disorders) | 7 (16)
Diarrhoea (Gastrointestinal disorders) | 9 (11)
Nausea (Gastrointestinal disorders) | 43 (149)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/14/NCT05246514/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/14/NCT05246514/SAP_001.pdf